CLINICAL TRIAL: NCT01086306
Title: Comparison of Risk of Hospitalization for Infections Between Patients With Type 2 Diabetes Exposed to Saxagliptin and Those Exposed to Other Oral Anti-Diabetic Treatments
Brief Title: Risk of Hospitalized Infections Among Patients With Type 2 Diabetes Exposed to Oral Antidiabetic Treatment
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: CV181-101
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients exposed to Saxagliptin
- Patients exposed to oral antidiabetic drugs (not Saxagliptin)

SUMMARY:
The purpose of this study is to compare the incidence of hospitalizations for infections among patients with type 2 diabetes mellitus who are new initiators of Saxagliptin and those who are new initiators of Oral Anti-Diabetic Drug (OADs) in classes other than DPP4 inhibitors; and to compare the incidence of hospitalizations with infections associated with T-lymphocyte dysfunction (i.e., herpes zoster, tuberculosis, or non-tuberculous mycobacterial infections [evaluated as a composite outcome]) among patients with type 2 diabetes mellitus who are new initiators of Saxagliptin and those who are new initiators of OADs in classes other than DPP4 inhibitors.

DETAILED DESCRIPTION:
Prospectively designed retrospective database study. This study will be conducted using administrative claims data and electronic medical records that are collected as part of routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Newly prescribed Saxagliptin [or an OAD in a class other than Dipeptidyl peptidase-4 (DPP4) inhibitors]
* Enrolled in the respective database for at least 180 days prior to the first prescription of new OAD

Exclusion Criteria:

* Patients identified with a diagnostic code for inpatient diagnostic code for any of the infections of interest within the 180-day baseline period
* Patients with DPP4 inhibitor exposure during the baseline period
* Patients currently using exenatide or insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out using databases containing administrative claims data [HealthCore Integrated Research Database (HIRD) and Medicare in the U.S.] and electronic medical records [General Practice Research Database (GPRD) and The Health Improvement Network (THIN) in the UK]. The US population includes patients from health plans in the northeast, southeastern, mid-Atlantic, central, mid-western, and western regions (HIRD) as well as US citizens 65 years of age and older (Medicare). The UK population includes patients seeking medical care from general practitioners (GPRD and THIN)
Sampling Method: Non-Probability Sample
Enrollment: 113505 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To compare the incidence of hospitalizations for infections among patients with type 2 Diabetes Mellitus who are new initiators of Saxagliptin and those who are new initiators of oral antidiabetic drug (OADs) in classes other than DPP4 inhibitors | 18 months
To compare the incidence of hospitalizations for infections among patients with type 2 Diabetes Mellitus who are new initiators of Saxagliptin and those who are new initiators of oral antidiabetic drug (OADs) in classes other than DPP4 inhibitors | 36 months
To compare the incidence of hospitalizations for infections among patients with type 2 Diabetes Mellitus who are new initiators of Saxagliptin and those who are new initiators of oral antidiabetic drug (OADs) in classes other than DPP4 inhibitors | 54 months
To compare the incidence of hospitalizations with infections associated with T Lymphocyte dysfunction | 18 months
  To compare the incidence of hospitalizations with infections associated with T Lymphocyte dysfunction (i.e., herpes zoster, tuberculosis, or non-tuberculous mycobacterial infections[evaluated as a composite outcome]) among patients with type 2 Diabetes Mellitus who are new initiators of Saxagliptin and those who are new initiators of OADs in classes other than DPP4 inhibitors
To compare the incidence of hospitalizations with infections associated with T Lymphocyte dysfunction | 36 months
  To compare the incidence of hospitalizations with infections associated with T Lymphocyte dysfunction (i.e., herpes zoster, tuberculosis, or non-tuberculous mycobacterial infections[evaluated as a composite outcome]) among patients with type 2 Diabetes Mellitus who are new initiators of Saxagliptin and those who are new initiators of OADs in classes other than DPP4 inhibitors
To compare the incidence of hospitalizations with infections associated with T Lymphocyte dysfunction | 54 months
  To compare the incidence of hospitalizations with infections associated with T Lymphocyte dysfunction (i.e., herpes zoster, tuberculosis, or non-tuberculous mycobacterial infections[evaluated as a composite outcome]) among patients with type 2 Diabetes Mellitus who are new initiators of Saxagliptin and those who are new initiators of OADs in classes other than DPP4 inhibitors

SECONDARY OUTCOMES:
A composite outcome of either inpatient or outpatient diagnoses of herpes zoster, tuberculosis, and non-tuberculous mycobacterial infections plus prescriptions for related antimicrobial therapies | 18 months
A composite outcome of either inpatient or outpatient diagnoses of herpes zoster, tuberculosis, and non-tuberculous mycobacterial infections plus prescriptions for related antimicrobial therapies | 36 months
A composite outcome of either inpatient or outpatient diagnoses of herpes zoster, tuberculosis, and non-tuberculous mycobacterial infections plus prescriptions for related antimicrobial therapies | 54 months
Inpatient or outpatient diagnoses of herpes zoster, tuberculosis, or non-tuberculous mycobacterial infections (evaluated separately) | 18 months
Inpatient or outpatient diagnoses of herpes zoster, tuberculosis, or non-tuberculous mycobacterial infections (evaluated separately) | 36 months
Inpatient or outpatient diagnoses of herpes zoster, tuberculosis, or non-tuberculous mycobacterial infections (evaluated separately) | 54 months
Inpatient diagnoses of respiratory tract infections | 18 months
Inpatient diagnoses of respiratory tract infections | 36 months
Inpatient diagnoses of respiratory tract infections | 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Lo Re V, Carbonari DM, Saine ME, Newcomb CW, Roy JA, Liu Q, Wu Q, Cardillo S, Haynes K, Kimmel SE, Reese PP, Margolis DJ, Apter AJ, Reddy KR, Hennessy S, Bhullar H, Gallagher AM, Esposito DB, Strom BL. Postauthorization safety study of the DPP-4 inhibitor saxagliptin: a large-scale multinational family of cohort studies of five outcomes. BMJ Open Diabetes Res Care. 2017 Jul 31;5(1):e000400. doi: 10.1136/bmjdrc-2017-000400. eCollection 2017. PMID 28878934
- [Derived] Saine ME, Carbonari DM, Newcomb CW, Nezamzadeh MS, Haynes K, Roy JA, Cardillo S, Hennessy S, Holick CN, Esposito DB, Gallagher AM, Bhullar H, Strom BL, Lo Re V 3rd. Determinants of saxagliptin use among patients with type 2 diabetes mellitus treated with oral anti-diabetic drugs. BMC Pharmacol Toxicol. 2015 Apr 2;16:8. doi: 10.1186/s40360-015-0007-z. PMID 25889498
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4450&filename=cv181_101.pdf